CLINICAL TRIAL: NCT01428011
Title: Racial Differences in Patient-Provider Communication and Medication Adherence
Brief Title: Patient-Provider Communication and Medication Adherence
Acronym: MEDCHAT
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-00311; 1K23HL098564-01A1 (NIH)
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
Keywords: Hypertension; Patient-Provider Communication; Medication Adherence; Race Concordance
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No treatment: African American/Black and Caucasian/White patients with hypertension

SUMMARY:
The purpose of this study is to understand how communication between African American and white patients with high blood pressure and his/her primary care provider effects whether a patient decides to take their high blood pressure medications.

DETAILED DESCRIPTION:
High blood pressure contributes to the racial disparities in death rates between minority patients and whites. Understanding the factors underlying racial disparities in high blood pressure-related outcomes is a major focus of Healthy People 2010. Several factors including access to care, patient preferences and lower socioeconomic status have been used to explain the differences seen in timely and effective delivery of preventive care between minority patients and whites. However, when these factors are controlled for, health disparities still exist. Recently, the Institute of Medicine identified interpersonal processes within the patient-provider relationship as a potential reason for the health disparities between minority and white patients. Specifically, providers' communication, including the ability to listen, collaborate, and be empathetic during the medical encounter has emerged as an important dimension of care that differs by race. Despite the increasing evidence that racial differences in patient-provider communication affects patient care, many of these studies have examined issues related to processes of care such as patient satisfaction with little attention to intermediate outcomes such as medication adherence. Further, studies that have used audio-taped analysis to examine racial differences in patient-provider communication are limited by one-dimensional coding systems that lack the ability to capture the mutual influence the patient and provider have on one another during the interaction. Thus, the potential pathways through which patient-provider communication contribute to high blood pressure-related disparities in minority patients compared to whites is not clearly understood. This proposed two-phase, mixed-methods research study, provides a unique opportunity to address these gaps by clarifying the effect of patient's race on patient-provider communication and medication adherence among 120 hypertensive African American and white patients receiving care in primary care practices. Specifically, findings from a qualitative analysis of patient-provider communication (Phase 1) will inform the development of a conceptual model that will be used to quantitatively evaluate the relationship between patient's race, patient-provider communication and medication adherence (Phase 2).

ELIGIBILITY:
Inclusion Criteria:

* self-identification as black/African American or white/Caucasian
* Receiving care in the Bellevue Hospital Ambulatory Care Practice from the same primary care provider for at least 3 months;
* Diagnosed with hypertension (ICD: # 401-401.9)
* Taking at least one antihypertensive medication;
* Age18 years or older
* Fluent in English

Exclusion Criteria:

* Unable to give informed consent
* Refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from Primary Care Clinics in New York City
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | 3-months
  Medication adherence will be assessed as a continuous variable with the Medication Event Monitoring System (MEMS) and calculated as the percent of prescribed doses removed by the patient during the 3-month stud

SECONDARY OUTCOMES:
patient-provider communication | Baseline
  Patient-provider communication will be assessed with the validated Medical Interaction Process System (MIPS). Patient-provider communication will be defined as ratios using formulas derived from the audiotaped analysis. Ratios will be calculated by dividing the sum of all codes for the communication behavior of interest (e.g., provider dominated-talk) by the sum of all codes for the comparison communication behavior of interest (e.g., patient-dominated-talk).

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Schoenthaler, EdD, Principal Investigator — NYU School of Medicine
Locations (1):
- Bellevue Hospital Ambulatory Care Practive, New York, New York, United States